CLINICAL TRIAL: NCT00708253
Title: Single- vs. Double-balloon Enteroscopy in Small Bowel Diagnostics: A Randomized Controlled Single-blind Multicenter Trial
Brief Title: Single- Versus Double-balloon Enteroscopy in Small Bowel Diagnostics
Acronym: SBE_vs_DBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: University Hospital Muenster, Dept. of Medicine B
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SBE-DBE_2008
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Gastrointestinal Diseases
Keywords: balloon assisted enteroscopy; single balloon enteroscopy; double balloon enteroscopy; insertion depth
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SBE (Active Comparator)
  Interventions: Device: Single-balloon procedure (SBE)
- DBE (Active Comparator)
  Interventions: Device: Double-balloon procedure (DBE)

INTERVENTIONS:
Device: Double-balloon procedure (DBE) — Double-balloon procedure (DBE): DBE is performed using the DBE T-type endoscope system (Fujinon Inc, Japan), as described in the literature. The DBE endoscope consist of a 200-cm long video endoscope with an outer diameter of 8.5 mm and a flexible overtube with a length of 145 cm and an outer diameter of 12 mm. Latex balloons are attached to both the endoscope and the overtube. These balloons are inflated and deflated during insertion, as described elsewhere in detail (2,3).
  Arms: DBE
Device: Single-balloon procedure (SBE) — Single-balloon procedure (SBE): SBE is performed using the SBE endoscope system (SIF-Q180, Olympus Optical Co., Ltd., Tokyo, Japan). The SBE endoscope consist of a 200-cm long video endoscope with an outer diameter of 9.2 mm and a flexible overtube with a length of 140 cm and an outer diameter of 13.2 mm. One single balloon is attached to the the tip of the overtube. The insertion process follows the method used for DBE, but instead of inflation of the endoscope balloon, the tip of the endoscope is angulated at straightening
  Arms: SBE

SUMMARY:
Background: The small bowel has been a black box for gastrointestinal (GI) endoscopy as, until recently, most of the small bowel was not accessible with conventional endoscopes. Double-balloon enteroscopy (DBE) is an endoscopic procedure for visualizing the entire small bowel. The method was first described by Yamamoto and colleagues in 2001. Both endoscopic diagnosis and treatment can be easily performed using DBE. The first larger series, recently published, demonstrate that DBE is feasible in visualizing large parts of the small bowel. Although DBE has widely been used routinely for examining the small intestine there are a few issues which may limit its use. The preparation and handling of the DBE-endoscope is often interpreted as being complex (such as attaching the balloon to the tip of the endoscope, inflating/deflating the two balloon systems).

Recently, a novel balloon enteroscope system has been developed using only a single balloon (single balloon enteroscope, SBE). SBE was designed to facilitate diagnosis and treatment of the small bowel. The endoscopist needs to manipulate only one single balloon; thereby, time and complexity for preparation of the system and for the examination itself may be reduced. However, the new SBE system may be less efficient for deep intubation of the small bowel and may cause adverse effects due to the hooking of the endoscope during straightening of the endoscope.

Study Aim: The primary aim of the present study is to compare the new SBE system with the standard DBE system with respect to completeness of visualisation and insertion depth of the small bowel, as well as complications during the procedure.

DETAILED DESCRIPTION:
Study design:

The study is designed as a multicenter randomized controlled trial. The participating centers are Rikshospitalet University Hospital (Dept. of Gastroenterology), Oslo, Norway, University Hospital Muenster (Dept. of Medicine B), Muenster, Germany and Erasmus Medical Center, Rotterdam, The Netherlands.

Randomization:

Randomization to SBE or DBE is performed on basis of the individual participant. Equally large groups are randomized using block randomization (blocks of six patients) for each of the participating centers. Randomization (using SPSS statistical software package) is performed by an independent researcher, who is not part of the endoscopy team.

Double-balloon procedure:

DBE is performed using the DBE T-type endoscope system (Fujinon Inc, Japan), as described in the literature. The DBE endoscope consist of a 200-cm long video endoscope with an outer diameter of 8.5 mm and a flexible overtube with a length of 145 cm and an outer diameter of 12 mm. Latex balloons are attached to both the endoscope and the overtube. These balloons are inflated and deflated during insertion, as described elsewhere in detail.

Single-balloon procedure:

SBE is performed using the SBE endoscope system (SIF-Q180, Olympus Optical Co., Ltd., Tokyo, Japan). The SBE endoscope consist of a 200-cm long video endoscope with an outer diameter of 9.2 mm and a flexible overtube with a length of 140 cm and an outer diameter of 13.2 mm. One single balloon is attached to the the tip of the overtube. The insertion process follows the method used for DBE, but instead of inflation of the endoscope balloon, the tip of the endoscope is angulated at straightening.

Ethics:

The regional ethics committees of the participating centers will be asked for approval of the study protocol.

Power analysis:

The present study is a non-inferiority study, aiming on showing equality between the two endoscope systems with regard to the main endpoints. A pilot study including 20 patients in each group will be performed since there is no data in present literature with respect to the main endpoints. The difference in percentage of complete visualization between the two groups will be used as the power-driving endpoint. The results of the pilot study will then be used for power calculation of the study applying the no inferiority-thesis. P-values of < 0.05 will be considered statistically significant.

Ad addendum:

The manufacturer of one of the instruments on the present trial (Olympus) approached the investigators in late January 2009 about a possible risk of increased adverse events with the Olympus endoscope. The company was not aware of any details regarding the nature of these events or the magnitude of this potential risk, as the warning was solely based on unpublished rumors in the GI community. To prevent participants in the present trial from any harm, the investigators decided to perform an interim analysis including all patients included in the trial until February 1, 2009, to rule out possible adverse events or poor performance in one or both of the involved treatment arms. No stopping rules apply for this interim analysis.

ELIGIBILITY:
Inclusion criteria:

* Patients referred for routine balloon enteroscopy where total enteroscopy is indicated
* All individuals provide written informed consent before entering the trial

Exclusion criteria:

* Age under 18 years
* Inability to understand information for participation
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Comparison of completeness of visualization of the small bowel by combination of upper and lower balloon enteroscopy | 12 months

SECONDARY OUTCOMES:
Comparison of small bowel insertion depth, time to complete visualization of the small bowel (combined approaches), patient discomfort, use of sedatives during the procedure, diagnostic yield, complications and adverse effects due to the procedure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Domagk, M.D., Principal Investigator — University of Muenster, Dept. of Medicine B; Lars Aabakken, M.D., Principal Investigator — Rikshospitalet University Hospital, Dept. of Medicine; Peter Mensink, M.D., Principal Investigator — Erasmus University Medical Center, Dept. of Gastroenterology and Hepatology; Michael Bretthauer, M.D., PhD, Study Chair — Rikshospitalet University Hospital, Dept. of Medicine
Locations (3):
- University of Muenster, Dept. of Medicine B, Münster, Germany
- Erasmus University Medical Center, Dept. of Gastroenterology and Hepatology, Rotterdam, Netherlands
- Rikshospitalet University Hospital, Dept. of Medicine, Oslo, Norway

REFERENCES:
- [Background] Yamamoto H, Sekine Y, Sato Y, Higashizawa T, Miyata T, Iino S, Ido K, Sugano K. Total enteroscopy with a nonsurgical steerable double-balloon method. Gastrointest Endosc. 2001 Feb;53(2):216-20. doi: 10.1067/mge.2001.112181. PMID 11174299
- [Background] Ell C, May A, Nachbar L, Cellier C, Landi B, di Caro S, Gasbarrini A. Push-and-pull enteroscopy in the small bowel using the double-balloon technique: results of a prospective European multicenter study. Endoscopy. 2005 Jul;37(7):613-6. doi: 10.1055/s-2005-870126. PMID 16010603
- [Background] May A, Nachbar L, Ell C. Double-balloon enteroscopy (push-and-pull enteroscopy) of the small bowel: feasibility and diagnostic and therapeutic yield in patients with suspected small bowel disease. Gastrointest Endosc. 2005 Jul;62(1):62-70. doi: 10.1016/s0016-5107(05)01586-5. PMID 15990821
- [Background] Domagk D, Bretthauer M, Lenz P, Aabakken L, Ullerich H, Maaser C, Domschke W, Kucharzik T. Carbon dioxide insufflation improves intubation depth in double-balloon enteroscopy: a randomized, controlled, double-blind trial. Endoscopy. 2007 Dec;39(12):1064-7. doi: 10.1055/s-2007-966990. PMID 18072057
- [Background] Hartmann D, Eickhoff A, Tamm R, Riemann JF. Balloon-assisted enteroscopy using a single-balloon technique. Endoscopy. 2007 Feb;39 Suppl 1:E276. doi: 10.1055/s-2007-966616. Epub 2007 Oct 24. No abstract available. PMID 17957636
- [Background] Tsujikawa T, Saitoh Y, Andoh A, Imaeda H, Hata K, Minematsu H, Senoh K, Hayafuji K, Ogawa A, Nakahara T, Sasaki M, Fujiyama Y. Novel single-balloon enteroscopy for diagnosis and treatment of the small intestine: preliminary experiences. Endoscopy. 2008 Jan;40(1):11-5. doi: 10.1055/s-2007-966976. Epub 2007 Dec 4. PMID 18058613
- [Result] Maaser C, Ullerich H, Menzel K, Domagk D, Lügering A, Domschke W, Kucharzik T. Double balloon enteroscopy - a useful diagnostic tool? Analysis of a large, non-selected cohort of patients regarding success and complication of double-balloon endoscopy (abstract). Gastroenterology 2006;130:A476.